CLINICAL TRIAL: NCT04409899
Title: The Utility of Enhanced Pre- and Post-surgical Protocols to Prevent the Spread of COVID-19 in a Large Urological Department (UroCovid Study)
Brief Title: The Utility of Enhanced Pre and Post-surgical Work-out to Prevent the Spread of COVID-19 in a Large Urology Department
Acronym: UroCovid
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fundacio Puigvert (Other)
Responsible Party: Principal Investigator, Francesco Sanguedolce, MD, PhD, FEBU, Fundacio Puigvert
Other Study IDs: FundacióPuigvert
Record Dates: First submitted 2020-05-26; First posted 2020-06-01 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: COVID-19; Urologic Diseases; Surgery--Complications; Epidemic Disease
Keywords: Pre-surgical screening; Post-surgical work out; Urological surgery; Nosocomial COVID-19 incidence
MeSH Terms: conditions — COVID-19; Urologic Diseases | interventions — Hematologic Tests; COVID-19 Nucleic Acid Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Urological surgical patients during COVID-19 pandemic: During the COVID-19 pandemic, the urological patients in the need of a surgical intervention have been screened on the basis of the underline conditions, the priority of surgery, and risk-benefit assessment. A pre-surgical work-out was performed in the selected patients, with some of them being detected of COVID-19 at RT-PCR or suspected for it according to the risk-assessment survey. Enhanced blood tests and X-rays of the thorax were performed as baseline assessments. In case of development of post-surgical unspecific symptoms, clinical and laboratory work-out were performed before to expedite a new RT-PCR, which would have required preventive isolation of a patient in a COVID-19 ward. We evaluated the impact of COVID-19 in this selected cohort and the complications eventually associated with the viral infection.
  Interventions: Diagnostic Test: Blood tests

INTERVENTIONS:
Diagnostic Test: Blood tests — RT-PCR, D-dimer, CRP, procalcitonin, ferritin, complete haemogram
  Other Names: RT-PCR

SUMMARY:
Since the outbreak of COVID-19 hit Spain in March 2020, most of the elective surgeries have been canceled everywhere. As soon as the epidemiology phase of the pandemic changed and the restrictions have been eased, different protocols have been put in place to screen patients for SARS-CoV-2 before surgery in order to reduce the spreading of the disease in hospitalized patients. To the best of the current state of knowledge, no recommendations or protocols have been established to guide surgeons in dealing with patients developing unspecific symptoms after surgeries, which could sign either of a post-op complication or COVID-19. The investigators have developed an enhanced pre and post-surgical protocol both to screen patients for COVID-19 before surgery and to promptly identify those patients suspicious for the viral infection during the post-op.

DETAILED DESCRIPTION:
The pandemic outbreak of SARS-CoV-2 has put significant strain on the hospitals of many countries around the world. Spain has been one of the countries most affected by the COVID-19, with nearly 30 thousands of confirmed deaths as by 23rd of May 2020.

While the state of emergency was declared by the Spanish government at the beginning of March 2020, the Intensive Care Units of the larger Spanish cities were overwhelmed by the number of patients in need of invasive respiratory supports. Moreover, data from China revealed that patients undergoing surgery and being SARS-CoV-2 carriers were at higher risk for complications and fatalities. As a result, most of the elective surgeries have been canceled in all surgical disciplines. As far as it concerned the urology patients, recommendations were provided by the European Association of Urology in order to guide the selection of the surgeries to be prioritized. Further recommendations on how to screen patients before surgeries were released by other national and international scientific societies and regulatory boards.

However, regardless of a successful pre-operative screening with patients being cleared of COVID-19, there might be still the possibility the patients could incubate the virus during hospitalization or getting it in the hospital from other patients, visitors or professionals.

To the best of the current state of knowledge, no recommendations have been published on how to guide the decision-making process on patients developing postoperatively unspecific symptoms (fever, chest pain, oxygen desaturation, etc) which could raise suspicions for COVID-19 during the outbreak of the disease.

The Institutional site of the investigators is a monographic hospital fully dedicated to urology and nephrology, and work in close cooperation with one of the four larger public hospitals in Barcelona; this latter has been one of those hospitals under significant strain for the COVID-19 emergency, while the former was marginally involved by the pandemic wave. The urological surgical activities never stopped during the outbreak, though initially were severely reduced; after experiencing some post-operative severe complications in patients developing concomitantly the SARS-CoV-2 infection, the investigators developed an enhanced pre and post-surgical protocol having a twofold objective: 1) to limit the risk to intervene patients harbouring the SARS-CoV-2 by undertaking an RT-PCR test 48 hours before surgery, and screening for symptoms compatible with COVID-19 and/or for strict contacts with infected people; furthermore, an X-ray thorax, and serum D-dimer and C-Reactive Protein were undertaken to establish baseline values. 2) to establish a post-surgical algorithm to guide surgeons on the nature of unspecific (and common) symptoms that could overlook for COVID-19 or rather raise unnecessary alarms for the viral infection, by performing serum/blood and imaging tests.

As soon as the protocol was put in action, data have been recorded prospectively in a registry in order to evaluate the utility of such a strategy. The recruitment period has been planned to embrace only the acute phase of the pandemic; the investigators hypothesize that such enhanced work-out may reduce the hospital contamination and optimal patient care in the acute phase of the COVID-19 pandemic as well as in its future waves, especially in those urological or surgical sites where activities have not been discontinued.

ELIGIBILITY:
Inclusion Criteria:

* Patients selected for urological surgery during COVID-19 pandemic

Exclusion Criteria:

* Patients admitted in the hospital not undergoing surgical intervention

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in a waiting list for a urological surgery and selected to undertake the intervention during COVID-19 pandemic according to priority and risk/benefit assessment
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of SARS-CoV-2/COVID-19 in a selected cohort of urological patients undergoing surgery | Day 1 pre-op up to day-30 post-op
Post-operative COVID-19 related complication rates | Day 1 pre-op up to day-30 post-op

SECONDARY OUTCOMES:
Association between post-surgery inflammatory indexes and COVID-19 diagnosis during hospitalization | Up to day-30 post-op

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Sanguedolce, MD, PhD, Principal Investigator — Fundacio Puigvert
Locations (1):
- Fundacio Puigvert, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
At the moment there is no plan to share data, but it could be considered in case of need

REFERENCES:
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Shang W, Dong J, Ren Y, Tian M, Li W, Hu J, Li Y. The value of clinical parameters in predicting the severity of COVID-19. J Med Virol. 2020 Oct;92(10):2188-2192. doi: 10.1002/jmv.26031. Epub 2020 Jun 2. PMID 32436996
- [Background] Lippi G, Plebani M. Procalcitonin in patients with severe coronavirus disease 2019 (COVID-19): A meta-analysis. Clin Chim Acta. 2020 Jun;505:190-191. doi: 10.1016/j.cca.2020.03.004. Epub 2020 Mar 4. No abstract available. PMID 32145275
- [Background] Stensland KD, Morgan TM, Moinzadeh A, Lee CT, Briganti A, Catto JWF, Canes D. Considerations in the Triage of Urologic Surgeries During the COVID-19 Pandemic. Eur Urol. 2020 Jun;77(6):663-666. doi: 10.1016/j.eururo.2020.03.027. Epub 2020 Apr 9. PMID 32279903
- [Background] Lei S, Jiang F, Su W, Chen C, Chen J, Mei W, Zhan LY, Jia Y, Zhang L, Liu D, Xia ZY, Xia Z. Clinical characteristics and outcomes of patients undergoing surgeries during the incubation period of COVID-19 infection. EClinicalMedicine. 2020 Apr 5;21:100331. doi: 10.1016/j.eclinm.2020.100331. eCollection 2020 Apr. PMID 32292899
- See also: World Health Organization. COVID-19 Situation Report — http://www.who.int/emergencies/diseases/novel-coronavirus-2019/situation-reports/